CLINICAL TRIAL: NCT02903758
Title: Frequency and Distribution of Mixed Falciparum-vivax Infections in French Guiana
Acronym: MixMal
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: universite de guyane (Unknown)
Responsible Party: Sponsor
Other Study IDs: mixmalaria
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Cross-Sectional Studies

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — malaria parasites
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cross sectional

SUMMARY:
Malaria is still endemic in the interior of French Guiana. mixed infections by 2 or more different malaria parasites lead to complex and potentially harmfull therapeutic problems. The aim of the study was to look at malaria smears between 2000 and 2008 and determine using PCR the frequency of mixed infections, and their distribution in the terrtory of French Guiana. Overall 10.75% of 400 smears showed mixed infection with P. falciparum and P. vivax. The Maroni river where Duffy negative populations live was largely devoid of vivax infections. These results suggest that mixed infections are frequent in french guiana except on the Maroni river which leads to practical implications for clinicians facing a patient with clinical malaria.

ELIGIBILITY:
Inclusion Criteria:

* malaria diagnosis

Exclusion Criteria:

* no malaria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: malaria positive patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2000-01; Primary Completion 2000-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
malaria | At the time of diagnosis of malaria
  PCR positive for malaria parasites

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana, France

IPD SHARING:
Plan to Share IPD: No